# **Application Form of Buddhist Tzu Chi Medical Foundation**"Clinical Research on Jingsi Bencao Decoction"

| Application number | • |
|--------------------|---|
| 1 1 | |

| <b>A</b> | | • | • 4 | • | | • | |
|-------------------------------|----|-----|-----|-----|-------|-----|---|
| <b>A.</b> | Ka | 212 | int | Ori | m ๑ 1 | חוד | n |
| $\boldsymbol{\Omega} \bullet$ | Da | 210 | | ULI | ma | UU | ш |

sign in person)
Signature and seal of the co-host of

the project (please

| 7 X D | asic illioi | mation | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Plan | Chinese | 淨斯本草飲 | 濃縮 | 夜對長新 | 冠症狀- | 腸腦軸失 | 調之身 | 中心症狀 | 療效-隨機等 | 雙盲臨床試驗 |
| name Jing Si Herbal Tea Liquid Packet in the treatment of psychophysical burden in patients with disorders of long-COVI double-blind, randomized, placebo-controlled study | | | | | | | | | | |
| Inve | incipal<br>estigator<br>Name | Chen,<br>Chien-Lin | Job<br>title | | ctor of<br>nterology | Campus | <u>Huali</u><br>Chi H | ien Tzu<br>Iospital | unit<br>or<br>department | Gastroenterology |
| | execution<br>period | ■One year<br>From Jan | nuary | 1, 2012 to | o Decem | ber 31, 20 | 012, a t | otal of 1 | year. | |
| case. (C<br>■ Yes, p | o-hosted pro<br>project name: | jects will not<br>Exploring th | be cone rela | unted)<br>itionship | between | supragas | tric bel | ching, pł | nysical and | spital, a total of 1<br>mental symptoms,<br>I reflux disease. |
| | r the project | has carried o | out the | followin | ng related | l experim | ents: [] | f von tic | k any of the | e following items, |
| | 1 3 | e relevant ex | | | $\boldsymbol{\mathcal{C}}$ | | | ir you tre | on any or an | e rome wing nems, |
| _ | a to attach th | c relevant ex | рстип | JIII/ICSCAI | ich consc | iii docuii | icitsj | | | |
| □ No. | | | | <i></i> | | | | | | 11. |
| ■ Huma | n experimen | ts/human spe | cımen | is (includ | ing huma | an embryo | | - | | ells).<br>nust be attached. |
| Progra | am Contact | 姓名: <u>Cher</u><br>E-MAIL: <u>h</u> | | _ | - | | | | | ) 0988-282055 |
| Signati | are and seal | | | | | | | | | |
| _ | host of the | | | | | | | | | |
| | total | | | | , Date | : Y | <i>l</i> ear | Mon | th Da | av |
| | lease sign in | | | | _ | | | | | 3 |
| | erson) | | | | | | | | | |
| | are and seal | | | | | | | | | |
| | co-host of | | | | , Date | | loor | Mon | th D | 24.7 |
| the pro | ject (please | | | | _ , Date | 1 | lear | Mon | thDa | 1y |
| sign i | in person) | | | | | | | | | |
| Signati | are and seal | | | | | | | | | |
| | co-host of | | | | , Date | : Y | /ear | Mon | th Da | av. |
| | ject (please | | | | | 1 | · • | 1V1011 | D | * <i>y</i> |
| ) | in person) | | | | | | | | | |
| _ | are and seal | | | | | | | | | |
| | co-host of | | | | , Date | : \ | <i>Y</i> ear | Mon | th Da | av |
| the pro | ject (please | | | | | · | | | | - <del>-</del> J |

, Date:\_\_\_\_Year\_\_\_

| sign in person) | | | | |
|---|---|---|---|---|
| Signature and seal<br>of the co-host of<br>the project (please<br>sign in person) | , Date: | Year | Month | Day |
| Dean's signature (personal signature or seal) | <br>, Date: | Year | Month | Day |

Remarks: If there are more than one co-hosts of the plan, please add the column by yourself to facilitate signature

# B. Personnel participating in the plan

| Category (moderator, co-host, co-host, researcher, etc.) | Name | Current position | The specific nature, project and scope of work undertaken in this research project |
|---|---|---|---|
| Moderator | Chen,<br>Chien-Lin | Director of Gastroenterology | Project progress supervision, research conduct and research plan formulation, data analysis analysis and report writing. |
| Co-host | Wong,<br>Ming-Wun | Attending Physician of Gastroenterology | Actual case acceptance, case processing, and data collation in the plan. |
| Co-host | Liu, Tso-Tsai | Director of<br>Endoscopy<br>Department | Actual case acceptance, case processing, and data collation in the plan. |
| Co-host | Yi,<br>Chih-Hsun | Attending Physician of Gastroenterology | Actual case acceptance, case processing, and data collation in the plan. |
| Co-host | Lei, Wei-Yi | • | Actual case acceptance, case processing, and data collation in the plan. |
| Co-host | Hung,<br>Jui-Sheng | | Actual case acceptance, case processing, and data collation in the plan. |
| Co-host | Liang,<br>Shu-Wei | Attending Physician of Gastroenterology | Actual case acceptance, case processing, and data collation in the plan. |
| Co-host | Liu,<br>Chin-Hung | Associate Professor | Specimen analysis, data analysis and statistics in the plan. |
| Co-host | Chen,<br>Chun-Yao | Assistant professor | Specimen analysis, data analysis and statistics in the plan. |

| Research assistant | Jian,<br>Yu-Xhuan | Research assistant | Organize data, data analysis and statistics and handle administrative affairs. |
|---|---|---|---|
|---|---|---|---|

**XIf** there are not enough fields, please copy by yourself.

## C. Implementation of other research projects

In the past three years, the project host, co-hosts, and other research team members must fill in the details of the implementation of the research plan.

| Category (moderator, co-host, co-host, researcher, etc.) | Name | Project name | Jobs<br>within the<br>plan | from year to<br>month | Grant agencies |
|---|---|---|---|---|---|
| Host | Chen,<br>Chien-Lin | To explore the pathophysiological effects of esophageal contraction, mucosal integrity and acid sensitivity on gastroesophageal reflux disease and the basis for treatment strategies | Host | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Host | Chen,<br>Chien-Lin | Efficacy of Jingsi Bencao Decoction on physical and mental symptoms of functional dyspepsia-a randomized double-blind clinical trial | Host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Host | Chen,<br>Chien-Lin | Discuss the pathophysiological mechanism of gastroesophageal reflux disease and establish the basis for accurate diagnosis and treatment based on esophageal reflux clearance ability, mucosal integrity and physical and mental characteristics | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Chen,<br>Chien-Lin | Discussion on the Pathophysiological Mechanism of Laryngopharyngeal Reflux Disease: Clinical Application of Artificial Intelligence Assisted and Accurate Diagnosis and Personalized Treatment Strategies | Co-host | 2022/8/1~<br>2025/07/31 | Ministry of<br>Science and<br>Technology |
| Host | Chen,<br>Chien-Lin | Discuss the pathophysiological mechanism and treatment strategy of afferent nerve distribution, esophageal peristalsis and drug regulation in gastroesophageal reflux disease | Co-host | 2022/8/1~<br>2025/07/31 | Ministry of<br>Science and<br>Technology |
| Host | Chen,<br>Chien-Lin | To explore the influence and clinical application of opioid analgesics on the pathophysiological mechanism of esophageal contraction and reflux characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Chen,<br>Chien-Lin | Analysis of 24-hour esophageal acid-base impedance | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |

| Version date: | (Version 3, | | | | |
|---|---|---|---|---|---|
| | | examination-technical | | | |
| | | performance and clinical | | | |
| | | application of gastroesophageal | | | |
| | | reflux disease diagnosis with | | | |
| | | artificial intelligence of | | | |
| | | supervised learning | | | |
| | | Application of high-resolution | | | |
| | | impedance pharyngeal function | | | |
| Host | Chen, | test and Sydney swallowing | Co-host | 2022/1/1~ | Hualien Tzu |
| поѕі | Chien-Lin | , | Co-nost | 2022/12/31 | Chi Hospital |
| | | questionnaire in oropharyngeal | | | |
| | | dysphagia and voice disorders | | | |
| | | Application of artificial | | | |
| | | intelligence in high-resolution | | | |
| Host | Chen, | esophageal function examination | Co-host | 2022/1/1~ | Hualien Tzu |
| 1103t | Chien-Lin | - research on unsupervised | Co-nost | 2022/12/31 | Chi Hospital |
| | | algorithm model based on deep | | | |
| | | learning | | | |
| | | To explore the influence of | | | |
| | | clinical characteristics and | | | |
| | Chen, | intestinal flora in patients with | ~ . | 2022/1/1~ | Hualien Tzu<br>Chi Hospital |
| Host | Chien-Lin | metabolism-related fatty liver | Co-host | 2022/12/31 | |
| | | under the regulation of diet and | | 2022/12/31 | Cin Trospitar |
| | | exercise | | | |
| | | To explore the role of esophageal | | | |
| | Chen,<br>Chien-Lin | | | | |
| 114 | | microbiota in novel impedance | Uost | 2021/1/1~ | Hualien Tzu |
| Host | | parameters, clinical classification | Host | 2021/12/31 | Chi Hospital |
| | | and hypersensitivity in | | | 1 |
| | | gastroesophageal reflux disease | | | |
| | | Clinical application of new | | | |
| | | esophageal impedance basic | Host | | |
| Host | Chen,<br>Chien-Lin | value supplemented with risk | | 2020/1/1~<br>2020/12/31 | Hualien Tzu |
| 1103t | | assessment to predict treatment | | | Chi Hospital |
| | | response and recurrence of | | | |
| | | gastroesophageal reflux disease | | | |
| | | To explore the relationship | | | |
| | | between esophageal acid | | | |
| | ~- | sensitivity, second-degree | | | |
| Co-host | Chen, | contraction of esophagus and | Co-host | 2021/1/1~ | Hualien Tzu |
| Co nost | Chien-Lin | subtypes of gastroesophageal | ee nest | 2021/12/31 | Chi Hospital |
| | | reflux and the pathogenic | | | |
| | | mechanism | | | |
| | | Clinical Application of | | | |
| | | High-resolution Impedance | | | |
| C - 1 4 | Chen, | 1 | C - 1 4 | 2021/1/1~ | Hualien Tzu |
| Co-host | Chien-Lin | Pharyngeal Function Examination | Co-host | 2021/12/31 | Chi Hospital |
| | | in Investigating Pharyngeal | | | 1 |
| | | Dysphagia and Drug Response | | | |
| Co-host | Chen, | Can a cure for hepatitis C | Co-host | 2020/1/1~ | Hualien Tzu |
| 20 11051 | Chien-Lin | improve quality of life? | 20 11050 | 2020/12/31 | Chi Hospital |
| | Chen, | Improving the quality of fatty | | 2020/1/1~ | Hualien Tzu |
| Co-host | Chien-Lin | liver treatment with cross-group | Co-host | 2020/1/1~<br>2020/12/31 | |
| | Cincii-Lin | care | | ZUZU/1Z/31 | Chi Hospital |
| | Cl | Discussion of differences in drug | | 2020/1/1 | II 1' T |
| Co-host | Chen, | therapy in patients with sensitive | Co-host | 2020/1/1~ | Hualien Tzu |
| 123 | Chien-Lin | esophagus and the role of | ~~- | 2020/12/31 | Chi Hospital |
| | <u>l</u> | | | | ı |

| Version date | (version 3, | | | | 1 |
|---|---|---|---|---|---|
| | | mucosal afferent innervation in | | | |
| | | this disease | | | |
| Co-host | Chen,<br>Chien-Lin | To explore the pathophysiological role of esophageal mucosal afferent nerve distribution in gastroesophageal reflux disease complicated with esophageal motility dysfunction | Co-host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Co-host | Chen,<br>Chien-Lin | Improve the diagnosis of laryngopharyngeal reflux disease and establish the indication of hydrogen ion pump blocker by using the average basic mucosal impedance value of the proximal esophagus at night | Co-host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Host | Wong,<br>Ming-Wun | Discussion on the Pathophysiological Mechanism of Laryngopharyngeal Reflux Disease: Clinical Application of Artificial Intelligence Assisted and Accurate Diagnosis and Personalized Treatment Strategies | Host | 2022/8/1~<br>2025/07/31 | Ministry of<br>Science and<br>Technology |
| Host | Wong,<br>Ming-Wun | Analysis of 24-hour esophageal acid-base impedance examination-technical performance and clinical application of gastroesophageal reflux disease diagnosis with artificial intelligence of supervised learning | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | Discuss the pathophysiological mechanism of gastroesophageal reflux disease and establish the basis for accurate diagnosis and treatment based on esophageal reflux clearance ability, mucosal integrity and physical and mental characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | To explore the influence and clinical application of opioid analgesics on the pathophysiological mechanism of esophageal contraction and reflux characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | Application of high-resolution impedance pharyngeal function test and Sydney swallowing questionnaire in oropharyngeal dysphagia and voice disorders | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | Application of artificial intelligence in high-resolution esophageal function examination - research on unsupervised algorithm model based on deep | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |

| version date | (Version 3, | 11/10/2022) | | | |
|---|---|---|---|---|---|
| | | learning | | | |
| Host | Wong,<br>Ming-Wun | To explore the influence of clinical characteristics and intestinal flora in patients with metabolism-related fatty liver under the regulation of diet and exercise | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | Efficacy of Jingsi Bencao Decoction on physical and mental symptoms of functional dyspepsia-a randomized double-blind clinical trial | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Host | Wong,<br>Ming-Wun | Improve the diagnosis of laryngopharyngeal reflux disease and establish the indication of hydrogen ion pump blocker by using the average basic mucosal impedance value of the proximal esophagus at night | Host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Host | Wong,<br>Ming-Wun | To explore the role of esophageal microbiota in novel impedance parameters, clinical classification and hypersensitivity in gastroesophageal reflux disease | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | To explore the relationship<br>between esophageal acid<br>sensitivity, second-degree<br>contraction of esophagus and<br>subtypes of gastroesophageal<br>reflux and the pathogenic<br>mechanism | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | Clinical Application of High-resolution Impedance Pharyngeal Function Examination in Investigating Pharyngeal Dysphagia and Drug Response | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | To explore the pathophysiological effects of esophageal contraction, mucosal integrity and acid sensitivity on gastroesophageal reflux disease and the basis for treatment strategies | Co-host | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Host | Wong,<br>Ming-Wun | Can a cure for hepatitis C improve quality of life? | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | Improving the quality of fatty liver treatment with cross-group care | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |
| Host | Wong,<br>Ming-Wun | Clinical application of new esophageal impedance basic value supplemented with risk assessment to predict treatment response and recurrence of gastroesophageal reflux disease | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |

| version date | (version 3, | 11/10/2022) | | <u></u> | _ |
|---|---|---|---|---|---|
| Host | Wong,<br>Ming-Wun | Discussion of differences in drug<br>therapy in patients with sensitive<br>esophagus and the role of<br>mucosal afferent innervation in<br>this disease | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Yi,<br>Chih-Hsun | Exploring the relationship between esophageal contraction, esophageal mucosal integrity and esophageal mucosal afferent nerves: the mechanism of influence on esophageal dysfunction and gastroesophageal reflux | Co-host | 2017/8/1~<br>2020/07/31 | Ministry of<br>Science and<br>Technology |
| Co-host | Liu,<br>Tso-Tsai | To explore the influence of clinical characteristics and intestinal flora in patients with metabolism-related fatty liver under the regulation of diet and exercise | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liu,<br>Tso-Tsai | Discuss the pathophysiological mechanism of gastroesophageal reflux disease and establish the basis for accurate diagnosis and treatment based on esophageal reflux clearance ability, mucosal integrity and physical and mental characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liu,<br>Tso-Tsai | To explore the influence and clinical application of opioid analgesics on the pathophysiological mechanism of esophageal contraction and reflux characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liu,<br>Tso-Tsai | Application of high-resolution impedance pharyngeal function test and Sydney swallowing questionnaire in oropharyngeal dysphagia and voice disorders | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liu,<br>Tso-Tsai | Analysis of 24-hour esophageal acid-base impedance examination-technical performance and clinical application of gastroesophageal reflux disease diagnosis with artificial intelligence of supervised learning | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liu,<br>Tso-Tsai | Application of artificial intelligence in high-resolution esophageal function examination - research on unsupervised algorithm model based on deep learning | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liu,<br>Tso-Tsai | Efficacy of Jingsi Bencao<br>Decoction on physical and mental | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical |

| Version date | (Version 3, | | | | |
|---|---|---|---|---|---|
| | | symptoms of functional | | | Corporation |
| | | dyspepsia-a randomized | | | |
| | | double-blind clinical trial | | | |
| | | To explore the role of esophageal | | | |
| | | microbiota in novel impedance | | | |
| Co-host | Liu, | parameters, clinical classification | Co-host | 2021/1/1~ | Hualien Tzu |
| Co nost | Tso-Tsai | and hypersensitivity in | Co nost | 2021/12/31 | Chi Hospital |
| | | gastroesophageal reflux disease | | | |
| | | To explore the relationship | | | |
| | | between esophageal acid | | | |
| | Liu, | sensitivity, second-degree | | 2021/1/1~ | Hualien Tzu |
| Co-host | Tso-Tsai | contraction of esophagus and | Co-host | 2021/12/31 | Chi Hospital |
| | 130 1341 | subtypes of gastroesophageal | | 2021/12/31 | Cin Hospitai |
| | | reflux and the pathogenic | | | |
| | | mechanism | | | |
| | | Clinical Application of | | | |
| | | High-resolution Impedance | | 2021/1/1 | 11 1: m |
| Co-host | Liu, | Pharyngeal Function Examination | Co-host | 2021/1/1~ | Hualien Tzu |
| 00 11050 | Tso-Tsai | in Investigating Pharyngeal | 00 11000 | 2021/12/31 | Chi Hospital |
| | | Dysphagia and Drug Response | | | |
| | | Improving the quality of fatty | | | |
| Co-host | Liu, | liver treatment with cross-group | Host | 2020/1/1~ | Hualien Tzu |
| Co-nost | Tso-Tsai | | поя | 2020/12/31 | Chi Hospital |
| | τ. | care | | 2020/1/1 | 11 1: T |
| Co-host | Liu, | Can a cure for hepatitis C | Co-host | 2020/1/1~ | Hualien Tzu |
| | Tso-Tsai | improve quality of life? | | 2020/12/31 | Chi Hospital |
| | | Clinical application of new | | | |
| | Liu,<br>Tso-Tsai | esophageal impedance basic | | 00001414 | |
| Co-host | | value supplemented with risk | Co-host | 2020/1/1~ | Hualien Tzu |
| Co-nost | | assessment to predict treatment | Co-nost | 2020/12/31 | Chi Hospital |
| | | response and recurrence of | | | _ |
| | | gastroesophageal reflux disease | | | |
| | | Discussion of differences in drug | | | |
| | | therapy in patients with sensitive | | | |
| Co-host | Liu, | esophagus and the role of | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu |
| Co nost | Tso-Tsai | mucosal afferent innervation in | | | Chi Hospital |
| | | this disease | | | |
| _ | | | | | |
| | | To explore the pathophysiological | | | |
| | τ. | effects of esophageal contraction, | | | Ministry of |
| Co-host | Liu, | mucosal integrity and acid | Co-host | 2020/8/1~ | Science and |
| | Tso-Tsai | sensitivity on gastroesophageal | | 2023/07/31 | Technology |
| | | reflux disease and the basis for | | | |
| | | treatment strategies | | | |
| | | Discuss the pathophysiological | | | |
| | | mechanism and treatment strategy | | | Ministry of |
| C - 1 4 | T -: XV-: X/: | of afferent nerve distribution, | TT4 | 2022/8/1~ | Ministry of |
| Co-host | Lei, Wei-Yi | esophageal peristalsis and drug | Host | 2025/07/31 | Science and |
| | | regulation in gastroesophageal | | | Technology |
| | | reflux disease | | | |
| | | To explore the influence and | | | |
| | | clinical application of opioid | | | |
| Co-host | | analgesics on the | | 2022/1/1~ | Hualien Tzu |
| | Lei, Wei-Yi | | Host | 2022/1/1~ 2022/12/31 | |
| | | pathophysiological mechanism of | | 2022/12/31 | Chi Hospital |
| | | esophageal contraction and reflux | | | |
| | | characteristics | | | |

| Version date | · (version 3, | 11/10/2022) | | | |
|---|---|---|---|---|---|
| Co-host | Lei, Wei-Yi | Discuss the pathophysiological mechanism of gastroesophageal reflux disease and establish the basis for accurate diagnosis and treatment based on esophageal reflux clearance ability, mucosal integrity and physical and mental characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Lei, Wei-Yi | Application of high-resolution impedance pharyngeal function test and Sydney swallowing questionnaire in oropharyngeal dysphagia and voice disorders | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Lei, Wei-Yi | Application of artificial intelligence in high-resolution esophageal function examination - research on unsupervised algorithm model based on deep learning | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Lei, Wei-Yi | Analysis of 24-hour esophageal acid-base impedance examination-technical performance and clinical application of gastroesophageal reflux disease diagnosis with artificial intelligence of supervised learning | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Lei, Wei-Yi | To explore the influence of clinical characteristics and intestinal flora in patients with | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Lei, Wei-Yi | dyspepsia-a randomized<br>double-blind clinical trial | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Co-host | Lei, Wei-Yi | To explore the pathophysiological role of esophageal mucosal afferent nerve distribution in gastroesophageal reflux disease complicated with esophageal motility dysfunction | Host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Co-host | Lei, Wei-Yi | and hypersensitivity in gastroesophageal reflux disease | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Lei, Wei-Yi | To explore the relationship<br>between esophageal acid<br>sensitivity, second-degree<br>contraction of esophagus and<br>subtypes of gastroesophageal | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |

| TOTOTION date | (version 5, | | I | | |
|---|---|---|---|---|---|
| | | reflux and the pathogenic mechanism | | | |
| | | Clinical Application of | | | |
| 0.1.4 | 1 . 337 . 37. | High-resolution Impedance | C 1 4 | 2021/1/1~ | Hualien Tzu |
| Co-host | Lei, Wei-Yi | Pharyngeal Function Examination | Co-host | 2021/1/~ 2020/1/1~ 2020/12/31 2020/12/31 2020/12/31 2020/12/31 2020/12/31 2020/12/31 2020/12/31 2020/8/1~ 2023/07/31 2017/8/1~ 2020/07/31 2022/12/31 2022/12/31 | Chi Hospital |
| | | in Investigating Pharyngeal | | | 1 |
| | | Dysphagia and Drug Response | | | |
| Co-host | Lei, Wei-Yi | Can a cure for hepatitis C | Co-host | | Hualien Tzu |
| | 201, 1101 11 | improve quality of fife? | 00 11000 | 2020/12/31 | Chi Hospital |
| | | Improving the quality of fatty | | 2020/1/1~ | Hualien Tzu |
| Co-host | Lei, Wei-Yi | liver treatment with cross-group | Co-host | | Chi Hospital |
| | | care | | 2020/12/31 | CIII 1105pittii |
| | | Clinical application of new | | | |
| | | esophageal impedance basic | | | |
| Co-host | Lei, Wei-Yi | value supplemented with risk | Co-host | 2020/1/1~ | Hualien Tzu |
| Co-nost | Lei, Wei-11 | assessment to predict treatment | Co-nost | 2020/12/31 | Chi Hospital |
| | | response and recurrence of | | | |
| | | gastroesophageal reflux disease | | | |
| | | Discussion of differences in drug | | | |
| | | therapy in patients with sensitive | | 2020/1/1 | H1: T |
| Co-host | Lei, Wei-Yi | | Host | | Hualien Tzu |
| | | mucosal afferent innervation in | | 2020/12/31 | Chi Hospital |
| | | this disease | | | |
| | | To explore the pathophysiological | | | |
| | | effects of esophageal contraction, | | 2020/12/31<br>2020/8/1~<br>2023/07/31 | 25. |
| ~ . | | mucosal integrity and acid | | | Ministry of |
| Co-host | Lei, Wei-Yi | sensitivity on gastroesophageal | Co-host | | Science and |
| | | reflux disease and the basis for | | | Technology |
| | | treatment strategies | | | |
| | | Exploring the relationship | | 2020/12/31<br>2020/12/31<br>2020/8/1~<br>2023/07/31<br>2017/8/1~<br>2020/07/31 | |
| | | between esophageal contraction, | | | |
| | | esophageal mucosal integrity and | | | |
| G 1 | | asonhagaal mucosal affarant | | | Ministry of |
| Co-host | Lei, Wei-Yi | nerves: the mechanism of | Co-host | | Science and |
| | | influence on esophageal | | 2020/07/01 | Technology |
| | | dysfunction and gastroesophageal | | | |
| | | reflux | | | |
| | | Application of high-resolution | | | |
| | | impedance pharyngeal function | | | |
| Co-host | Hung, | test and Sydney swallowing | Host | | Hualien Tzu |
| Co nost | Jui-Sheng | questionnaire in oropharyngeal | 1103t | 2020/12/31 2020/12/31 2020/8/1~ 2023/07/31 2017/8/1~ 2020/07/31 | Chi Hospital |
| | | dysphagia and voice disorders | | | |
| | | Discuss the pathophysiological | | | |
| | | mechanism of gastroesophageal | | | |
| | | reflux disease and establish the | | | |
| | Нипа | basis for accurate diagnosis and | | 2022/1/1- | Hualien Tzu |
| Co-host | Hung, Jui-Sheng | treatment based on esophageal | Co-host | | Chi Hospital |
| | Jui-Silcing | reflux clearance ability, mucosal | | 2022/12/31 | Cin Hospital |
| | | • | | | |
| | | integrity and physical and mental characteristics | | | |
| | T T | To explore the influence and | | 2022/1/1 | II1:- T |
| Co-host | Hung, | clinical application of opioid | Co-host | | Hualien Tzu |
| | Jui-Sheng | analgesics on the | | 2022/12/31 | Chi Hospital |
| | | pathophysiological mechanism of | | | |

| VOI BION GATO | | aconhaced contraction and reflux | | | |
|---|---|---|---|---|---|
| | | esophageal contraction and reflux characteristics | | | |
| Co-host | Hung,<br>Jui-Sheng | Analysis of 24-hour esophageal acid-base impedance examination-technical performance and clinical application of gastroesophageal reflux disease diagnosis with artificial intelligence of supervised learning | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | Application of artificial intelligence in high-resolution esophageal function examination - research on unsupervised algorithm model based on deep learning | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | To explore the influence of clinical characteristics and intestinal flora in patients with metabolism-related fatty liver under the regulation of diet and exercise | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | Efficacy of Jingsi Bencao Decoction on physical and mental symptoms of functional dyspepsia-a randomized double-blind clinical trial | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Co-host | Hung,<br>Jui-Sheng | Clinical Application of High-resolution Impedance Pharyngeal Function Examination in Investigating Pharyngeal Dysphagia and Drug Response | Host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | To explore the role of esophageal microbiota in novel impedance parameters, clinical classification and hypersensitivity in gastroesophageal reflux disease | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | To explore the relationship<br>between esophageal acid<br>sensitivity, second-degree<br>contraction of esophagus and<br>subtypes of gastroesophageal<br>reflux and the pathogenic<br>mechanism | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | Can a cure for hepatitis C improve quality of life? | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | Improving the quality of fatty liver treatment with cross-group care | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | Clinical application of new esophageal impedance basic value supplemented with risk assessment to predict treatment response and recurrence of | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |

| Version date: | (Version 3, | - | | | |
|---|---|---|---|---|---|
| | | gastroesophageal reflux disease | | | |
| Co-host | Hung,<br>Jui-Sheng | Discussion of differences in drug<br>therapy in patients with sensitive<br>esophagus and the role of<br>mucosal afferent innervation in<br>this disease | Co-host | 2020/1/1~<br>2020/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Hung,<br>Jui-Sheng | Discussion of differences in drug<br>therapy in patients with sensitive<br>esophagus and the role of<br>mucosal afferent innervation in<br>this disease | Co-host | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Co-host | Liang,<br>Shu-Wei | Application of artificial intelligence in high-resolution esophageal function examination - research on unsupervised algorithm model based on deep learning | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liang,<br>Shu-Wei | Analysis of 24-hour esophageal acid-base impedance examination-technical performance and clinical application of gastroesophageal reflux disease diagnosis with artificial intelligence of supervised learning | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liang,<br>Shu-Wei | Discuss the pathophysiological mechanism of gastroesophageal reflux disease and establish the basis for accurate diagnosis and treatment based on esophageal reflux clearance ability, mucosal integrity and physical and mental characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liang,<br>Shu-Wei | To explore the influence and clinical application of opioid analgesics on the pathophysiological mechanism of esophageal contraction and reflux characteristics | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liang,<br>Shu-Wei | To explore the influence of clinical characteristics and intestinal flora in patients with metabolism-related fatty liver under the regulation of diet and exercise | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Co-host | Liang,<br>Shu-Wei | Efficacy of Jingsi Bencao Decoction on physical and mental symptoms of functional dyspepsia-a randomized double-blind clinical trial | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Co-host | Liang,<br>Shu-Wei | To explore the role of esophageal microbiota in novel impedance parameters, clinical classification | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |

| Version date | : (Version 3, | 11/10/2022) | | | |
|---|---|---|---|---|---|
| | | and hypersensitivity in | | | |
| | | gastroesophageal reflux disease | | | |
| | | To explore the relationship | | | |
| | | between esophageal acid | | | |
| | Liona | sensitivity, second-degree | | 2021/1/1~<br>2021/12/31<br>2021/12/31<br>2020/08/01~<br>2022/07/31<br>2022/07/31<br>2022/12/31<br>2021/01/01~<br>2021/12/31<br>2019/10/01~<br>2020/09/30 | Hualien Tzu |
| Co-host | Liang,<br>Shu-Wei | contraction of esophagus and | Co-host | | Chi Hospital |
| | Silu- Wei | subtypes of gastroesophageal | | 2021/12/31 | Cili Hospitai |
| | | reflux and the pathogenic | | | |
| | | mechanism | | | |
| | | Clinical Application of | | | |
| | Liang, | High-resolution Impedance | | 2021/1/1- | Hualien Tzu |
| Co-host | Shu-Wei | Pharyngeal Function Examination | Co-host | | Chi Hospital |
| | Silu- WCI | in Investigating Pharyngeal | | 2021/12/31 | Cili Hospitai |
| | | Dysphagia and Drug Response | | | |
| | | Using bee indicators and | | | |
| | Liu, | geographic information system to | | 2020/08/01~ | Ministry of |
| Co-host | Chin-Hung | assess pesticide exposure in | Co-host | | Science and |
| | Cilli-Trung | different crops | | 2022/07/31 | Technology |
| | | MOST109-2314-B-320-002-MY2 | | | |
| | Liu, | Exploring the relationship | | 2021/12/31 2021/12/31 2020/08/01~ 2022/07/31 2022/01/01~ 2022/12/31 2021/101/01~ 2021/12/31 2019/10/01~ 2020/09/30 | |
| | | between cholesterol metabolism | | | |
| Co-host | Chin-Hung | pathway and drug insensitivity in | Host | | 慈濟大學 |
| | Cilli Trung | oral squamous cell carcinoma | | 2022/12/31 | |
| | | TCMRC-P-110011 | | | |
| | | Synergistic antitumor effects of | | | |
| | | statins and SREBP2 inhibitors in | | | |
| Co-host | Liu, | oral squamous cell carcinoma: the | Host | | 慈濟大學 |
| ee nost | Chin-Hung | role of the mevalonate pathway | 1103t | | 13.777 |
| | | and statin-insensitive features | | | |
| | | TCMRC-P-109009 | | | |
| | | Molecular mechanisms of statins | | | |
| | | inhibiting the growth of oral | | | |
| | Liu, | squamous cell carcinoma: the role | ** | 2019/10/01~ | 4 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| Co-host | Chin-Hung | of DNA methyltransferases and | Host | | 慈濟大學 |
| | | the regulation of turnor | | | |
| | | suppressor gene epigenetics | | | |
| | | TCMRC-P-108003 | | | |
| | | To explore the influence of | | | |
| | CI | clinical characteristics and | | | TT 1: T |
| Co-host | Chen, | intestinal flora in patients with | Co-host | | Hualien Tzu |
| | Chun-Yao | metabolism-related fatty liver | | 2022/12/31 | 2022/12/31 |
| | | under the regulation of diet and | | | |
| | | exercise | | | |

 $\mathbf{X}$  If there are not enough fields, please copy by yourself.

## **D.** Instructions for Expected Use of Funds(Funding will be included in the review

and scoring items, please do not make up)

- 1. Please provide a detailed description of the purpose and annual amount of each expense (including research labor costs, consumables, etc.), if the column is insufficient, please add it yourself.
- 2. Research manpower expenses shall not be diverted to other business expenses.

  [Funds for the first year] (Please copy the form yourself and list the estimated funds year by year)

  (New Taiwan dollars)

| project name | illustrate | unit price | quantity | total price |
|---|---|---|---|---|
| 1. Research manpower Full-time concurrently (Please refer to the regulations in the Medical Special Management Measures for relevant insurance premiums) | Full-time staff: (the second year of full-time assistant at the bachelor level) The highest rank of personnel is limited to the ninth level of master's degree, and the items included in the work remuneration, labor and health insurance employer-borne expenses, labor retirement employer-borne expenses and year-end bonuses are handled in accordance with the regulations of the implementing agency (up to 1.5 months as the upper limit). Subtotal | 32,240<br>2,689<br>37<br>1,632<br>1,998 | 13<br>12<br>12<br>12<br>12<br>12 | 419,120<br>32,268<br>444<br>19,584<br>23,976 |
| 2. Consumables, items and miscellaneous expenses | Computer peripheral consumables: printer ribbon, toner cartridge, ink cartridge, printer photosensitive drum/roller, special printing paper, etc. Miscellaneous: postage and telecommunications fees, printing fees, photocopying paper, photocopying fees, binding fees, stationery fees, poster production fees, computer data statistics fees, computer data analysis fees, paper submission fees, paper publication fees, etc. | 14,608<br>10,000 | | 14,608<br>10,000 |
| 3. Medicine expenses (Jingsi herbal drink concentrate, please fill in the quantity) | Subtotal Jingsi herbal drink concentrate (2 packs*30 days*150 people) Placebo (2 packs*30 days*150 people) Subtotal | 0 | 9,000<br>9,000 | 24,608<br>0<br>0 |
| 4. Subject subsidy | Subject allowance (subsidy) Subtotal | 1,200 | 150 | 180,000 |
| 5. Inspection fee<br>(Please fill in the<br>inspection items and<br>fees) | LC-MS sample processing and analysis, intestinal bacteria analysis Subtotal | 5,000 | 150 | 750,000<br>750,000 |
| | | | total | 1,450,000 |

## E. Summary of the plan in Chinese

Please give an overview of the main points of this project within 500 words, and customize keywords according to the nature of this project, and please write in Chinese.

新冠肺炎患者在痊癒後,約10%患者產生長新冠症狀,長新冠症狀中的腹痛、腹脹、腹瀉及便祕源自於腸腦軸失調,腸腦軸失調包含功能性消化不良和腸躁症,常規檢查無明顯異常,由於原因不明但盛行率高,往往對患者的身心健康影響甚鉅。即使腸腦軸失調目前被認為和胃腸道局部發炎和微生物菌相改變有關,但目前西醫治療療效不佳。有鑑於此,許多研究應用中草藥在功能性消化不良,並且達到不錯的療效。淨斯本草飲濃縮液為取得衛福部外銷專用許可證之食品,其成分為艾葉、魚針草、麥門冬、魚腥草、桔梗、甘草、紫蘇葉、菊花等臺灣本土八種能清潤、散寒、宣肺化痰、利濕清熱的中藥草,在臨床試驗登記立案作為輔助新冠肺炎的治療,目前初步發現亦可改善患者腸胃症狀以及憂焦慮程度。故本研究採雙盲隨機試驗,以淨斯本草飲濃縮液用於客觀檢查皆正常之長新冠症狀-腸腦軸失調患者,評估其治療前後之身心症狀以及腸道菌代謝產物之變化。

關鍵詞:長新冠症狀、腸腦軸失調、淨斯本草飲濃縮液、身心症狀

計畫概述:請概述執行本計畫之目的及可能產生對社會、經濟、學術發展等 面向的預期影響性(三百字以內)。

腸腦軸失調(DGBI)包含功能性消化不良和腸躁症為新冠肺炎感染後的腸胃 道問題,也是傳統西醫療效值得改善的疾病,淨斯本草飲濃縮液為東部地區 研發之中草藥食品,期待淨斯本草飲濃縮液在感染新冠肺炎病毒後改善腸胃 道功能以及憂鬱情況的發現能夠用於改善腸腦軸失調(DGBI)之身心症狀。

※此部分內容於獲核定補助後將逕予公開

**XIf** there are not enough fields, please copy by yourself.

## F. Summary of the plan in English

Please provide an overview of the main points of this project within 500 words, and customize keywords according to the nature of this project, and please write in English.

Dyspepsia refers to chronic or recurrent upper gastrointestinal symptoms. According to the Rome IV criteria, functional dyspepsia (FD) symptoms included meal-related fullness, early satiation, epigastric pain or burning which are unexplained after routine investigation. FD causes substantial psychophysical burden because of its unknown etiology and high prevalence. Although FD is currently associated with local inflammation of the gastrointestinal tract and microbiota alteration, current available treatments for FD are of limited effectiveness. In view of this, many studies have applied Chinese herbal medicine in FD and achieved some therapeutic benefit. The Jing Si Herbal Tea Liquid Packet composed of eight native Taiwanese herbs (wormwood, hickory grass, Ophiopogon japonicus, houttuynia cordata, platycodon, licorice, perilla leaves, chrysanthemum) has obtained a special export license from the Ministry of Health and Welfare. The Jing Si Herbal Tea Liquid Packet also has been registered in clinical trials as a complementary treatment for COVID-19. The preliminary data demonstrated that the Jing Si Herbal Tea Liquid Packet may improve gastrointestinal symptoms and anxiety in patients with COVID-19. Therefore, this study aims to investigate the impact of the Jing Si Herbal Tea Liquid Packet on psychophysical burden and metabolites of microbiota in patients with FD through a double-blind randomized manner.

關鍵詞: functional dyspepsia; Jing Si Herbal Tea Liquid Packet; psychophysical burden

**XIf there are not enough fields, please copy by yourself.** 

## G. Background and purpose of the research project

Please describe in detail the background, purpose, importance of this research project and the research situation related to this project at home and abroad,

Comments on important references, etc., please write in Chinese format.

#### **Background**

#### Symptoms of the new crown-gut-brain axis disorder (disorders of gut-brain interaction, DGBI)

COVID-19 is raging all over the world. The novel coronavirus recognizes type 2 angiotensin-converting enzyme and infects various cells in the body, including cells in the gastrointestinal tract. About 12%–20% of patients are infected and develop gastrointestinal symptoms. (1, 2) About 10% of patients with COVID-19 will develop symptoms of COVID-19 after recovery, (3) Abdominal pain, bloating, diarrhea and constipation in symptoms of COVID-19 originate from disorders of gut-brain interaction, DGBI). (4) In the upper gastrointestinal tract (upper abdominal pain, abdominal distension), it is called functional dyspepsia, and in the lower gastrointestinal tract (abdominal pain, diarrhea, constipation), it is called irritable bowel syndrome. (5) In a large-scale survey in the United States (more than 100,000 people), it was found that after the COVID-19 epidemic, the incidence of gut-brain axis disorder (DGBI) increased by 75% compared with before the epidemic. (6) Disorders of the gut-brain axis (DGBI) include functional dyspepsia and irritable bowel disorder. At present, there is no clear pathogenesis and standard treatment. The consensus is to use the Roman diagnostic criteria, evaluate by questionnaire, and exclude other organic diseases. disease to diagnose. (5) The possible mechanisms of gut-brain axis disorder (DGBI) include local inflammation of the gastrointestinal tract, infiltration and activation of allergic cells, mucosal defects, changes in microbial flora, and hypersensitivity of viscera. (7) In terms of the microbial flora of the brain-gut axis, the metabolites of intestinal bacteria are regarded as the key to influence, among which short-chain fatty acids (SCFA) are regarded as good metabolizers As a product, when carbohydrates are fermented, anaerobic bacteria will produce many short-chain fatty acids (SCFA) in the distal small intestine and colon, which are composed of 1-6 carbon atoms, and the main three metabolic compounds are acetic acid (Acetate), Propionate and Butyrate. Short-chain fatty acids (SCFA) have been shown in research to have anti-inflammatory, anti-oxidant, anti-diabetic, anti-cancer and antibacterial effects. When the bacterial phase changes, the concentration of short-chain fatty acids may change accordingly and affect human physiological responses. When the intestinal flora is out of balance, a variety of bad metabolites will be produced: Trimethylamine N-oxide, TMAO (derived from L-Carnitine or Choline), indoxyl sulfate (derived from Tryptophan) and p-cresyl sulfate (derived from Tyrosine), etc. (8)

#### Changes in the bacterial phase of the new crown symptoms

SARS-CoV-2 infection caused significant changes in the intestinal flora of patients. The number of

potential pathogens in the patient's body increases, and the antibiotic treatment also reduces the beneficial bacteria. <sup>9</sup> Hazan et al. (2022) showed reduced gut bacterial diversity in infected individuals, with reduced numbers of Bifidobacterium, Faecalibacterium, and Roseburium. <sup>10</sup> At six months post-infection, the intestinal bacterial diversity of the patients was still significantly low. <sup>11</sup> In addition to reduced diversity, these symptomatic patients had lower numbers of anti-inflammatory bacteria such as Faecalibacterium prausnitzii, Eubacterium rectale, Bifidobacterium adolescentis, and potential pathogens such as Rothia, Erysipelatoclostridium, Ruminococcus gnavus in the gut three months after infection. , Ruminococcus torques, and Bacteroides dorei are more. <sup>12</sup> Su et al. (2022) studied the dysbiosis caused by post-acute COVID-19 syndrome and found that there were more potential pathogens such as Erysipelatoclostridium ramosum and Ruminococcus gnavus, and beneficial bacteria Bifidobacterium adolescentis, B. pseudocatenulatum) decreased. <sup>13</sup> These evidences show that the intestinal flora has not fully recovered from the imbalance during infection, and is still in a state of low diversity and favorable pathogens, which can continue to cause immune responses in the intestine. Functional dyspepsia is also thought to be caused by increased permeability of the intestinal wall of the small intestine, allowing intestinal microbial metabolites to infiltrate the tissues and activate the immune system. <sup>14</sup>

In both functional dyspepsia and irritable bowel disorder, there is marked dysbiosis in the gut. Bacterial changes in patients with functional dyspepsia include decreased numbers of Bacteroidetes (Prevotellaceae) and increased numbers of Proteobacteria, Firmicutes (Streptococcus and Clostridia) and Bifidobacteria. 15 Bacterial changes in IBD included increased Clostridia (increased Ruminococcus but decreased Faecalibacterium), increased Lactobacillus and Streptococcus within the phylum Firmicutes, increased Bacteroides, and decreased Bifidobacteria. 16 After synthesis, it can be seen that the changes in the gut-brain axis disorder are mainly due to the replacement of Bacteroidetes by Firmicutes, while the changes in the number of Proteobacteria and Bifidobacteria are inconsistent.

#### Jing Si Herbal Tea Liquid Packet

The ingredients of Jing Si Herbal Tea Liquid Packet are mugwort leaves, houttuynia cordata, Ophiopogon japonicus, Houttuynia cordata, Campanulaceae, licorice, perilla leaves, chrysanthemum and other eight native Taiwanese herbs that can clear away moisture, dispel cold, relieve lungs and resolve phlegm, and clear away dampness and heat. Chinese medicinal herb, current research has found that it can block the combination of the new coronavirus and cells, and can also reduce cell penetration and block the virus from penetrating cells, while targeting wild-type and mutant viruses D614G, B.1.1.7, 501Y.V2 Carrying out animal studies, it was found that Jing Si Herbal Tea Liquid Packet can reduce the ability of 60 to 70% of the virus to infect the upper respiratory tract, lung, heart, and intestine of mice and reduce the expression of FKBP51, a protein related to depression, by 40%. The effect of using Jing Si Herbal Tea Liquid Packet to help reduce the amount of virus and systemic anti-inflammatory effect in patients with COVID-19. (9) In our

ongoing clinical study, for functional dyspepsia (FD) patients, Jing Si Herbal Tea Liquid Packet can improve symptoms in 75% of patients, compared with only 33% of placebo.

#### Purpose

A double-blind randomized trial was conducted to investigate the improvement of Jingsi Bencao decoction concentrate on the physical and mental symptoms of gut-brain axis disorder (DGBI) and the changes in intestinal flora after COVID-19.

#### **Importance**

Gut-brain axis disorders (DGBI), including functional dyspepsia and irritable bowel syndrome, are gastrointestinal problems after COVID-19 infection. They are also diseases that are worthy of improvement in the efficacy of traditional Western medicine. The discovery that Jingsi Bencao Drink Concentrate improves gastrointestinal function and depression after infection with the new coronavirus can be used to improve the physical and mental symptoms of gut-brain axis disorder (DGBI).

**XIf** there are not enough fields, please copy by yourself.

## H. Research methods, steps and implementation progress

- 1. Please describe in detail the research methods and reasons used in this project.
- 2. Estimated possible difficulties and solutions.
- 3. If it is a continuous plan, the research progress report or primary data of the previous year should be attached at the same time.
- 4. Please write in Chinese format.

#### 1. Subject acceptance and exclusion conditions

This study is a prospective study, which is expected to last for one year. It is planned to recruit 150 subjects with gut-brain axis disorder (DGBI) three months after being infected with new coronary pneumonia: 75 of them Functional dyspepsia (FD) subjects and 75 irritable bowel syndrome (IBS) subjects.

#### **Subject inclusion conditions (Inclusion criteria)**

- 1. Age between 20-70 years old.
- 2. Those who meet the definition of functional dyspepsia (FD).

(Functional dyspepsia (FD) is chronic (once a week, lasting at least three months, at least six months before the first symptom) upper gastrointestinal symptoms (any of the following): postprandial abdominal distension, easy to feel full, Epigastric pain or burning sensation in the upper abdomen, and no symptoms of gastrointestinal bleeding or significant weight loss, no abnormality after upper gastrointestinal endoscopy).

3. Those who meet the definition of irritable bowel syndrome (IBS).

(Irritable bowel syndrome (IBS) is chronic (once a week, lasting for at least three months) lower gastrointestinal symptoms: abdominal pain combined with diarrhea or constipation, and no symptoms of gastrointestinal bleeding or significant weight loss, no abnormalities after colonoscopy).

4.Be conscious and willing to sign the subject's consent form.

#### **Subject Exclusions (Exclusion criteria)**

- 1. Abnormal liver and kidney function;
- 2. Abnormal blood tests and thyroid abnormalities;
- 3. Have received surgery on the digestive tract;
- 4. Abnormal upper gastrointestinal endoscopy;
- 5. Abnormal colonoscopy;
- 6. Antibiotics are being used for infectious diseases;
- 7. Pregnant or breastfeeding women;
- 8. Suffering from heart, liver, or kidney failure;
- 9. Physical weakness, allergies, asthenia and cold constitution and chronic diseases.

#### 2. Experimental process

150 subjects with gut-brain axis disorder (DGBI) three months after being infected with new coronary

pneumonia will be recruited in the outpatient department of gastroenterology, including 75 subjects with functional dyspepsia (FD) and 75 subjects with irritable bowel syndrome (IBS) ) subjects; qualified subjects will receive blood and feces sampling and complete physical and mental symptom assessment (sleep habits questionnaire, anxiety questionnaire, stress questionnaire, gastrointestinal symptoms questionnaire, and irritable bowel syndrome questionnaire) before treatment, and then according to the double-blind random allocation method, the computer generated garbled characters, and assigned Jing Si Herbal Tea Liquid Packet or placebo according to the coding sequence, and the research assistant gave Jing Si Herbal Tea Liquid Packet or placebo, Host and recipients None of the subjects knew what the content of the assignment was. The experimenters took Jing Si Herbal Tea Liquid Packet or placebo in the first month, and after the end of the month, they received blood and stool tests and complete physical and mental symptom assessment (sleep habits questionnaire, anxiety questionnaire, stress questionnaire), gastrointestinal symptom questionnaire, and irritable bowel syndrome questionnaire), the laboratory will conduct pre- and post-test analysis of LC-MS and intestinal bacteria, and then conduct a cross-test. The original placebo will take Jing Si Herbal Tea Liquid Packet in the second month, previously taking Jing Si Herbal Tea Liquid Packet will take a placebo in the second month, after the end of the second month, do the third complete physical and mental symptom assessment (sleep habits questionnaire, anxiety questionnaire, stress questionnaire, digestive tract Symptom Questionnaire, Irritable Bowel Disorder Questionnaire), the test is completed.

#### Research flow chart



#### 3. Questionnaire

The questionnaire items included sleep habits questionnaire, anxiety questionnaire, stress questionnaire, gastrointestinal symptoms questionnaire, and irritable bowel syndrome questionnaire. The details of the questionnaire are attached.

#### 4. Collection, preservation, transportation and DNA extraction of feces

Fix the collection box on the toilet lid, discharge fresh feces into the collection box, then screw the lid tightly and place it in a zipper bag within 4 hours or in a -4°C refrigerator within 24-48 hours Sent to the laboratory for sub-packaging, and then refrigerated in a -80°C refrigerator. Thaw when the DNA is extracted, the extraction process includes the following steps sample homogenization, cell lysis, non-DNA material removal and DNA purification.

#### 5.Gut micrtobiota sequencing and community analysis

In this study, 16S rDNA massively parallel sequencing will be used to analyze the composition of gut bacteria. 0.25 g of stool samples were pooled for DNA extraction with the QIAmp PowerFecal Kit (Qiagen, Hilden, Germany). The purified DNA was PCRed with primers for 341F and 805R to amplify the V3-V4 fragments of the 16S rRNA gene, and the barcode was sent to the manufacturer for library building. The Illumina MiSeq platform was used for next-generation pair-end sequencing. Sample 30000 reads. After the sequence obtained by the manufacturer was screened for high-quality fragments by Mothur and Usearch software, the bacterial phase composition and taxonomic status of each sample were calculated. The taxonomic status of each sequence was determined by comparing the Mothur software with the SILVA sequence database. The investigators will use Microbiome Analyst R and other suitable R programming language packages to perform cluster analysis and network analysis of bacterial composition.

#### 6.Stool and Blood LC-MS Analysis

#### I. Plasma sample collection and preparation:

Whole blood was collected in Vacutainer K2E-EDTA (BD Diagnostics, Franklin Lakes, NJ, USA) blood collection tubes. The collected whole blood samples were then transferred to 15 mL containing Ficoll-paque PLUS medium [whole blood (hall blood)/ Ficoll-paque PLUS medium = 4/3 (volume ratio v/v)] (GE Healthcare Life Sciences, Pittsburgh, PA, USA) and centrifuge (3000 rpm, 30 min) at room temperature. After centrifugation, the plasma (plasma) supernatant that was successfully layered was collected and distributed into sterilized 1.5 mL microcentrifuge tubes (eppendorf), and glacial acetic acid with a concentration of 1 N and a volume of 1% was added.) aqueous solution to prevent the degradation of the analyte in plasma. Plasma is stored in a freezer at -80oC, and the storage period does not exceed 1 year.

#### **II.Previous processing method of Lipophilic Substances**:

Thaw the plasma sample at room temperature for 10-20 minutes, then transfer 100 µL of plasma to a new 1.5 mL microcentrifuge tube. Add the internal standard (internal control, 13C-PA) first, then add methanol 3 times the volume of plasma for deproteinization, and let it stand at room temperature for about 15-20 minutes. Then centrifuge the rested microcentrifuge tube (3,000 rpm, 10 min, 4 °C), and transfer the supernatant to the corresponding small glass test tube. Move the glass test tubes to a nitrogen blowing system, dry the samples through a nitrogen flow, and then add 100 µL of chloroform (Chloroform) to each sample for redissolution. A filtration extraction system was set up, and solid phase extraction columns [Solid phase extraction (SPE) columns (Strata-X-C 33 µm polymeric strong cation 60 mg/3 mL, Phenomenex, Torrance, CA, USA)] were used for extraction. Add 1.0-1.5 mL of n-hexane (hexane) solution to the erected column to activate the column, and use a vacuum pump to pump positive pressure for about 20-30 seconds. Replace the glass test tubes that have been filled with n-hexane solution under the filter extraction system, and then add the samples to the activated column in sequence. Add 1.0-1.5 mL of ethyl acetate (ethyl acetate) for vacuum extraction for about 30-45 seconds, and transfer the sample extracted with ethyl acetate to a nitrogen blowing system to dry it. Redissolve the sample with 100 µL of methanol, and finally transfer the reconstituted sample to a liquid chromatography-mass spectrometer (LC-MS) vial equipped with insert, and prepare for analysis on the machine with an injection volume of 30 µL per needle.

#### III. Hydrophilic Substances before the processing method:

There are two extraction methods for such compounds, namely traditional methanol extraction (Traditional deproteinized extraction) and SLE column extraction (SLE column extraction). First, place the plasma sample at room temperature to thaw for about 10-20 minutes. After the thawing is complete, take 100 µL to a new 1.5 mL microcentrifuge tube (two tubes of 100 µL are required for each sample). Plasma samples were deproteinized by adding methanol at a volume ratio of 3 times or adding an equal volume of 50 mM sodium phosphate dibasic heptahydrate (Sodium phosphate dibasic heptahydrate) and evenly mixed. Set up the SLE column filtration system and sample test tube, put the sample mixed with 50 mM disodium hydrogen phosphate hydrate into the column, turn on the vacuum pump to filter and extract, wait for about 3 minutes, then add 1.2-1.5 mL of acetic acid Ethyl esters are used for dike flushing. In addition, for the methanol deproteinized group, after waiting for about 20 minutes, they were centrifuged (3,000 rpm, 10 min, 4 °C), and then the supernatant was taken out into the corresponding glass test tube. The samples with two different treatment methods were put into the nitrogen blowing system for drying and concentration. For the group undergoing deproteinization, add 300 µL of methanol to redissolve, and filter with MILLEX GP 0.45 µM PVDF filter (Millipore), and discharge the liquid into the LC-MS special sample bottle loaded with insert; For the group extracted by the column, 100 µL of methanol was added for back-dissolution and reconstitution, and it was put into the LC-MS special sample bottle loaded with insert, ready for analysis on the machine.

#### d. LC-MS Analysis Conditions (Liquid Chromatography Mass Spectrometer):

LC-MS condition I: Used to analyze Lipophilic Substances

LC-MS condition II: Used to analyze Hydrophilic Substances Substances)

**Table 1. LC-MS analysis conditions:** 

| | LC cond | ditions | |
|---|---|---|---|
| HPLC system | Waters Alliance e2695 | Injection volume | 30 μL |
| | 60.0 min (I) | | Phenomenex Luna |
| Runtime | 60.0 min (I)<br>18.0 min (II) | Column | C18(2) |
| | 18.0 11111 (11) | | (250 x 4.6 mm, 5 μm) |
| Flow rate | 0.6 mL/min (I) | Column temp | 35°C (I) |
| riow rate | 0.8 mL/min (II) | Column temp | 40°C (I) |
| | Condiction I (Lipo) | philic Substances) | |
| Mobile | phase A | | phase B |
| 60:40 Acetonitrile: | ldH <sub>2</sub> O with 9.2 mM | 90:10 Isopropanol:Ac | etonitrile with 9.2 mM |
| Ammonium acetate (N | H <sub>4</sub> CH <sub>3</sub> CO <sub>2</sub> ) (pH 8.85) | Ammonium aceta | ate (NH <sub>4</sub> CH <sub>3</sub> CO <sub>2</sub> ) |
| Time (min) | %A | %B | Curve |
| Initial | 85 | 15 | 6 |
| 8.0 | 70 | 30 | 6 |
| 10.0 | 52 | 48 | 6 |
| 44.0 | 18 | 82 | 6 |
| 46.0 | 1 | 99 | 6 |
| 48.0 | 1 | 99 | 6 |
| 48.4 | 85 | 15 | 6 |
| 60.0 | 85 | 15 | 6 |
| | Condiction II (Hydro | ophilic Substances) | |
| Mobile | | | phase B |
| 0.1% Formic acid | l in 99.9% ddH2O | 0.1% Formic acid | d in 99.9% MeOH |
| Time (min) | %A | %B | Curve |
| 0 | 95 | 5 | 6 |
| 14 | 30 | 70 | 6 |
| 16 | 30 | 70 | 6 |
| 18 | 50 | 50 | 6 |
| | MS cond | ditions | |
| Detector | Waters ACQUITY QD | | |
| Ionization mode | ESI Negative (I); ESI I | Negative and Positive (I | I) |
| Capillary voltage | Default (0.8 kV) | | |
| Probe temp | Default (600°C) | | |
| Cone voltage | 20V(I); 15V(II) | | |
| Sampling rate | 8 Hz | | |
| Full scan | | 00 m/z for Negative (I); 70-600 m/z for Negative or Positive | |
| SIR | See <b>Table 2</b> - "Molecu | lar Ions (m/z)" | |

#### e. Method validation:

Including Limits of detection, LOD and Limits of quantitation, LOQ, Calibration curve, Recovery, accuracy and precision, Intra-assay, accuracy and precision and Inter-assay precision and accuracy of each test substance.

Table 2. LC-MS analysis Standard List:

| Molecular ion | Ion source |
|---------------|------------|
| (m/z) | mode |

| Propionate (3:0) 57+153 (3NPH) ESI Negative | ersion date: (Version 3 | <mark>, 11/10/2022)</mark> | | |
|---|---|---|---|---|
| Propionate (3:0) 57+153 (3NPH) ESI Negative | Lipophilic Substances | | | |
| Butyrate (4:0) S/F153 (3NPH) ESI Negative | Showt Chain Fatty | Acetate (2:0) | 42.0+153 (3NPH) | ESI Negative |
| Palmitic acid, PA (16:0) 255.1 ESI Negative | • | Propionate (3:0) | 57+153 (3NPH) | ESI Negative |
| Stearic Acid, SA (18:0) 283.2 ESI Negative | acius (SCFAS) | | 72+153 (3NPH) | ESI Negative |
| Palmitoleic Acid, POA (16:1) 253.2 ESI Negative | | Palmitic acid, PA (16:0) | 255.1 | ESI Negative |
| Oleic Acid, OA (18:1) 281.2 ESI Negative | Long Chain | Stearic Acid, SA (18:0) | 283.2 | ESI Negative |
| Fatty acid esters of hydroxy fatty acids (FAHFAs) Palmitoleic Acid Ester of 9-Hydroxystearic Acid (9-POHSA) Oleic Acid Ester of 9-Hydroxystearic Acid (9-OAHSA) Internal standards [13C16] - Palmitic acid (IS1) Palmitic acid (IS1) Thernal standards L-Methionine (L-Met) S-adenosyl-L-methionine (SAM) S-adenosyl-L-homocysteine (SAH) Antioxidants Ascorbic acid (MMA) Nutrition index Acetyl-L-histidine (3-MH) Fatty acids carrier Fatty acids carrier Palmitoleic Acid Ester of 9-Hydroxystearic Acid (9-POHSA) S-35.5 ESI Negative Sell Ne | Fatty acids | Palmitoleic Acid, POA (16:1) | 253.2 | ESI Negative |
| Patty acid esters of hydroxy fatty acids (FAHFAs) 9-Hydroxystearic Acid (9-POHSA) 563.5 ESI Negative | | Oleic Acid, OA (18:1) | 281.2 | ESI Negative |
| P-Hydroxystearic Acid (9-POHSA) Oleic Acid Ester of 9-Hydroxystearic Acid (9-OAHSA) ESI Negative | Fatty anid astors of | Palmitoleic Acid Ester of | 525.5 | ESI Nagatiya |
| Selic Acid Ester of 9-Hydroxystearic Acid (9-OAHSA) 563.5 ESI Negative | | 9-Hydroxystearic Acid (9-POHSA) | 333.3 | ESI Negative |
| Sel Positive | | Oleic Acid Ester of | 563.5 | ESI Nagatiya |
| | (FAIIFAS) | | 303.3 | ESI Negative |
| | | | <del>,</del> | |
| L-Methionine (L-Met)150.1ESI PositiveS-adenosyl-L-methionine (SAM)399.0ESI PositiveS-adenosyl-L-homocysteine (SAH)385.0ESI PositiveL-Homocysteine (L-Hcy)136.1ESI PositiveMethylmalonic acid (MMA)117.1ESI NegativeNutrition indexAscorbic acid (AA)174.9ESI NegativeNutrition index3-Methyl-L-histidine (3-MH)170.0ESI NegativeEatty acids carrierL-Carnitine (L-Car)162.1ESI PositiveFatty acids carrierAcetyl-L-Carnitine (ALC)204.0ESI PositivePropionyl-L-Carnitine (PLC)218.0ESI PositiveNephrotoxinIndoxyl Sulfate (InS)211.9ESI NegativeD-Cresyl sulfate (pCS)187.0ESI NegativeInternal standards153.1ESI Positive | $[^{13}C_{16}]$ | - Palmitic acid (IS1) | 271.4 | ESI Negative |
| S-adenosyl-L-methionine (SAM)399.0ESI Positive $S$ -adenosyl- $L$ -homocysteine (SAH)385.0ESI Positive $L$ -Homocysteine ( $L$ -Hcy)136.1ESI PositiveMethylmalonic acid (MMA)117.1ESI NegativeAntioxidantsAscorbic acid (AA)174.9ESI NegativeNutrition index3-Methyl- $L$ -histidine (3-MH)170.0ESI Negative $L$ -Carnitine ( $L$ -Car)162.1ESI PositiveFatty acids carrierAcetyl- $L$ -Carnitine (ALC)204.0ESI Positive $L$ -Carnitine (PLC)218.0ESI Positive $L$ -Carnitine (PLC)218.0ESI Positive $L$ -Carnitine (PLC) $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine (PLC) $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine (PLC) $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine (PLC) $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine (PLC) $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine $L$ -Carnitine <td< th=""><th></th><th>Hydrophilic Substances</th><th></th><th></th></td<> | | Hydrophilic Substances | | |
| Methionine cycleS-adenosyl-L-homocysteine (SAH)385.0ESI Positive $L$ -Homocysteine ( $L$ -Hcy)136.1ESI PositiveMethylmalonic acid (MMA)117.1ESI NegativeAntioxidantsAscorbic acid (AA)174.9ESI NegativeNutrition index3-Methyl- $L$ -histidine (3-MH)170.0ESI Negative $L$ -Carnitine ( $L$ -Car)162.1ESI PositiveAcetyl- $L$ -Carnitine (ALC)204.0ESI PositivePropionyl- $L$ -Carnitine (PLC)218.0ESI PositiveNephrotoxinIndoxyl Sulfate (InS)211.9ESI Negative $p$ -Cresyl sulfate (pCS)187.0ESI NegativeInternal standardsInternal standardsd3- $L$ -Methionine (d3- $L$ -Met) (IS2)153.1ESI Positive | | <i>L</i> -Methionine ( <i>L</i> -Met) | 150.1 | ESI Positive |
| | | S-adenosyl-L-methionine (SAM) | 399.0 | ESI Positive |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Methionine cycle | Palmitic acid (IS1) 271.4 Hydrophilic Substances L-Methionine (L-Met) 150.1 S-adenosyl-L-methionine (SAM) 399.0 | ESI Positive | |
| AntioxidantsAscorbic acid (AA) $174.9$ ESI NegativeNutrition index3-Methyl-L-histidine (3-MH) $170.0$ ESI NegativeL-Carnitine (L-Car) $162.1$ ESI PositiveFatty acids carrierAcetyl-L-Carnitine (ALC) $204.0$ ESI PositivePropionyl-L-Carnitine (PLC) $218.0$ ESI PositiveNephrotoxinTrimethylamine N-oxide (TMAO) $76.0$ ESI PositiveIndoxyl Sulfate (InS) $211.9$ ESI Negative $p$ -Cresyl sulfate (pCS) $187.0$ ESI NegativeInternal standardsd3-L-Methionine (d3-L-Met) (IS2) $153.1$ ESI Positive | | <i>L</i> -Homocysteine ( <i>L</i> -Hcy) | 136.1 | ESI Positive |
| Nutrition index3-Methyl- $L$ -histidine (3-MH)170.0ESI NegativeFatty acids carrier $L$ -Carnitine (L-Car)162.1ESI PositiveAcetyl- $L$ -Carnitine (ALC)204.0ESI PositivePropionyl- $L$ -Carnitine (PLC)218.0ESI PositiveNephrotoxinTrimethylamine $N$ -oxide (TMAO)76.0ESI PositiveIndoxyl Sulfate (InS)211.9ESI Negative $p$ -Cresyl sulfate (pCS)187.0ESI NegativeInternal standardsd3- $L$ -Methionine (d3- $L$ -Met) (IS2)153.1ESI Positive | | Methylmalonic acid (MMA) | 117.1 | ESI Negative |
| L-Carnitine (L-Car)162.1ESI PositiveAcetyl-L-Carnitine (ALC)204.0ESI PositivePropionyl-L-Carnitine (PLC)218.0ESI PositiveTrimethylamine N-oxide (TMAO)76.0ESI PositiveIndoxyl Sulfate (InS)211.9ESI Negative $p$ -Cresyl sulfate (pCS)187.0ESI NegativeInternal standardsd3-L-Methionine (d3-L-Met) (IS2)153.1ESI Positive | Antioxidants | Ascorbic acid (AA) | 174.9 | ESI Negative |
| Fatty acids carrierAcetyl-L-Carnitine (ALC)204.0ESI PositivePropionyl-L-Carnitine (PLC)218.0ESI PositiveNephrotoxinTrimethylamine $N$ -oxide (TMAO)76.0ESI PositiveIndoxyl Sulfate (InS)211.9ESI Negative $p$ -Cresyl sulfate (pCS)187.0ESI NegativeInternal standardsd3- $L$ -Methionine (d3- $L$ -Met) (IS2)153.1ESI Positive | Nutrition index | 3-Methyl- <i>L</i> -histidine (3-MH) | 170.0 | ESI Negative |
| Propionyl- $L$ -Carnitine (PLC) 218.0 ESI Positive Trimethylamine $N$ -oxide (TMAO) 76.0 ESI Positive Nephrotoxin Indoxyl Sulfate (InS) 211.9 ESI Negative $p$ -Cresyl sulfate (pCS) 187.0 ESI Negative Internal standards d3- $L$ -Methionine (d3- $L$ -Met) (IS2) 153.1 ESI Positive | | <i>L</i> -Carnitine (L-Car) | 162.1 | ESI Positive |
| | Fatty acids carrier | Acetyl- <i>L</i> -Carnitine (ALC) | 204.0 | ESI Positive |
| NephrotoxinIndoxyl Sulfate (InS)211.9ESI Negative $p$ -Cresyl sulfate (pCS)187.0ESI NegativeInternal standardsd3- $L$ -Methionine (d3- $L$ -Met) (IS2)153.1ESI Positive | J | Propionyl- <i>L</i> -Carnitine (PLC) | 218.0 | ESI Positive |
| p-Cresyl sulfate (pCS) 187.0 ESI Negative Internal standards d3-L-Methionine (d3-L-Met) (IS2) 153.1 ESI Positive | | Trimethylamine <i>N</i> -oxide (TMAO) | 76.0 | ESI Positive |
| Internal standards d3-L-Methionine (d3-L-Met) (IS2) 153.1 ESI Positive | Nephrotoxin | Indoxyl Sulfate (InS) | 211.9 | ESI Negative |
| d3-L-Methionine (d3-L-Met) (IS2) 153.1 ESI Positive | | <i>p</i> -Cresyl sulfate (pCS) | 187.0 | ESI Negative |
| d9-Trimethylamine N-oxide (d9-TMAO) (IS3) 85.0 ESI Positive | | | | ESI Positive |
| | d9-Trimethylam | ine N-oxide (d9-TMAO) (IS3) | 85.0 | ESI Positive |

### 7.Jing Si Herbal Tea Liquid Packet

In this experiment, Jing Si Herbal Tea Liquid Packet was used. Its ingredients are eight kinds of native Taiwan species, such as mugwort leaves, hinoki, Ophiopogon japonicus, Houttuynia cordata, bellflower, licorice, perilla leaves, and chrysanthemum. Dampness-clearing and heat-clearing herbs, take Jing Si Herbal Tea Liquid Packet 15 ml once a day in the morning and evening.





#### 8. Statistical Analysis

Continuous variables were expressed as mean and standard deviation if they were normally distributed; if they were not normally distributed, they were expressed as median and interquartile range. The treatment effect is presented by the improvement percentage of the sleep habits questionnaire, depression questionnaire, anxiety questionnaire, stress questionnaire, gastrointestinal symptoms questionnaire, and irritable bowel syndrome questionnaire before and after treatment, and the curative effect of Jingsi Bencao Drink Concentrate and placebo is expressed as the chi-square by the improvement percentage Chi-squared test comparison, P value less than 0.05 was considered statistically significant difference, the statistical analysis software used was SPSS 19 for Windows (SPSS, Inc, Chicago, IL, USA).

#### 9. Sample Size Estimation

According to our ongoing research, it is estimated that the efficacy of Jing Si Herbal Tea Liquid Packet for functional dyspepsia (FD) is 75%, while the efficacy of placebo is 33.3%. It is estimated by  $\alpha$ -error 0.05;  $\beta$ -error 0.20, at least 100 subjects are required to be admitted, and taking into account that the subjects may withdraw and fail to complete the trial successfully, the estimated number of subjects admitted in this study is 150.

#### 10. Possible difficulties and solutions

**Possible difficulties:** According to our current research, the effect of placebo on functional dyspepsia (FD) can reach 33.3%, so if the investigators want to prove that Jing Si Herbal Tea Liquid Packet has a positive effect on patients with new coronary pneumonia three months after infection Gut-brain axis dysregulation (DGBI) had to be statistically significantly greater than placebo to have a significant effect.

**Solution:** This trial adopts a multi-faceted whole-person care model to evaluate the curative effect, not only the symptoms of gut-brain axis disorder (DGBI) three months after being infected with new coronary pneumonia, but also the assessment of physical and mental symptoms, stress, and intestinal flora. Confirm the effect of Jing Si Herbal Tea Liquid Packet on various aspects of gut-brain axis disorder (DGBI).

#### 11. References

- 1. Mao R, Qiu Y, He JS, et al. Manifestations and prognosis of gastrointestinal and liver involvement in 1. Mao R, Qiu Y, He JS, et al. Manifestations and prognosis of gastrointestinal and liver involvement in patients with COVID-19: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol 2020;5:667-678.
- 2. Cheung KS, Hung IFN, Chan PPY, et al. Gastrointestinal Manifestations of SARS-CoV-2 Infection and Virus Load in Fecal Samples From a Hong Kong Cohort: Systematic Review and Meta-analysis. Gastroenterology 2020;159:81-95.
- 3. Golla R, Vuyyuru SK, Kante B, et al. Disorders of gut-brain interaction in post-acute COVID-19 syndrome. Postgrad Med J 2022.
- 4. Schmulson M, Ghoshal UC, Barbara G. Managing the Inevitable Surge of Post-COVID-19 Functional Gastrointestinal Disorders. Am J Gastroenterol 2021;116:4-7.
- 5. Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology 2016:1262-1279.
- 6. Aloysius MM, Goyal H, Ali A, et al. S220 Cancer-Specific 5-Year Survival Following Endoscopic Polypectomy versus Surgery for Malignant Colorectal Polyps. 2021;116:S97-S98.
- 7. Margolis KG, Cryan JF, Mayer EA. The Microbiota-Gut-Brain Axis: From Motility to Mood. Gastroenterology 2021;160:1486-1501.
- 8. Fan Y, Pedersen O. Gut microbiota in human metabolic health and disease. Nat Rev Microbiol 2021;19:55-71.
- 9. Zuo T, Wu X, Wen W, et al. Gut Microbiome Alterations in COVID-19. Genomics Proteomics Bioinformatics 2021;19:679-688.
- 10. Hazan S, Stollman N, Bozkurt HS, et al. Lost microbes of COVID-19: Bifidobacterium, Faecalibacterium depletion and decreased microbiome diversity associated with SARS-CoV-2 infection severity. BMJ Open Gastroenterol 2022;9.
- 11. Chen Y, Gu S, Chen Y, et al. Six-month follow-up of gut microbiota richness in patients with COVID-19. Gut 2022;71:222-225.
- 12. Tian Y, Sun KY, Meng TQ, et al. Gut Microbiota May Not Be Fully Restored in Recovered COVID-19 Patients After 3-Month Recovery. Front Nutr 2021;8:638825.
- 13. Su Q, Lau RI, Liu Q, et al. Post-acute COVID-19 syndrome and gut dysbiosis linger beyond 1 year after SARS-CoV-2 clearance. Gut 2022:gutjnl-2022-328319.
- 14. Wauters L, Ceulemans M, Schol J, et al. The Role of Leaky Gut in Functional Dyspepsia. Front Neurosci 2022;16:851012.
- 15. Zhou L, Zeng Y, Zhang H, et al. The Role of Gastrointestinal Microbiota in Functional Dyspepsia: A Review. Front Physiol 2022;13:910568.
- 16. Mazzawi T. Gut Microbiota Manipulation in Irritable Bowel Syndrome. Microorganisms 2022;10.
- 17. Hsieh PC, Chao YC, Tsai KW, et al. Efficacy and Safety of Complementary Therapy With Jing Si Herbal Tea in Patients With Mild-To-Moderate COVID-19: A Prospective Cohort Study. Front Nutr 2022;9:832321.